CLINICAL TRIAL: NCT06923813
Title: Assessment of Nutrient Absorption in Enterally Fed Post-ICU Patients Using Bomb Calorimetry: do the Calories Stick
Brief Title: Assessment of Nutrient Absorption in Enterally Fed Post-intensive Care Unit Patients Using Bomb Calorimetry: do the Calories Stick
Acronym: STICKY
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitair Ziekenhuis Brussel (Other)
Collaborators: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: STICKY
Record Dates: First submitted 2025-03-28; First posted 2025-04-11 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Post-ICU Patients Fully Enterally Fed
Keywords: PEG tube; indirect calorimetry; nasogastric
MeSH Terms: interventions — Energy Metabolism

STUDY DESIGN:
Intervention Model Description: 20 post-ICU patients who are fully enterally fed (PEG- or nasogastric tube)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participants (Experimental): 20 post-ICU patients who are fully enterally fed (PEG- or nasogastric tube). Step-by-Step Process: Every time a patient is included, all steps (caloric intake measurement, stool sample collection, blending, freezing, and freeze drying) will be performed sequentially. Bomb Calorimetry can be conducted either systematicallyfor a few patients at a time or all at once after all samples have been collected.
  Interventions: Other: caloric intake measurement; Procedure: stool sample collection; Other: energy expenditure measurement

INTERVENTIONS:
Other: caloric intake measurement — Detailed daily tracking of the enteral feeding provided to each patient, inclusing the type and amount of nutritional formula administered. Apart from the enteral intake, supplemental calories provided by infusion (e.g. glucose) will be recorded to ensure accurate measurement of caloric intake.
Procedure: stool sample collection — * a nonabsorbable blue dye marker will be administered at the start and end of the stool collection period to precisely indentify the stool produced within a specific time frame.
  * stool will be collected for three days. Each sample will be collected, weighted and labeled with the date and time, then stored at -20°C.
  * only stool samples from the appearance of the first dye marker to the appearance of the second dye marker will be saved and analyzed.
  * bomb calorimetry preparation
    * blending and dilution: each stool sample will be put into a blender and mixed with an equal amount of water
    * freeze dying: the diluted stool will be placed into freeze-dye flasks and frozen at -20°C. The next day, the flasks will be placed into a freeze dryer for 48hours.
    * pellet formation: the freeze-dried samples will be formed into 1-gram pellets and stored until calorimetry
    * calorimetry analysis: the Parr 6200 isoperibol calorimeter will be used to measure the energy content of the stool pellets
Other: energy expenditure measurement — performing indirect calorimetry to measure the REE of each patient

SUMMARY:
This study focuses on understanding how well patients who have recovered from an ICU stay absorb nutrients when receiving enteral (tube) feeding. Proper nutrition is crucial for recovery, but we don't fully understand how efficiently enteral feeding works in ICU survivors. The study will use advanced techniques like bomb calorimetry to measure the energy content of stool, and indirect calorimetry to measure patients' resting energy expenditure (REE). This will help assess the effectiveness of enteral feeding in these patients, providing valuable information about their metabolic needs and nutritional status.

The study will also look into the environmental impact of enteral feeding, particularly food waste. By understanding how much of the nutrition is absorbed versus excreted, the study hopes to suggest more sustainable feeding practices and reduce unnecessary waste in hospitals.

Key Goals:

* Primary Goal: Measure how much energy from enteral feeding is absorbed by patients post-ICU by analyzing their stool and energy expenditure.
* Secondary Goal: Assess how enteral feeding can be made more sustainable, with less waste generated from unused nutritional products.

This research will help improve nutritional care for ICU patients, enhance recovery, and potentially lead to more environmentally friendly healthcare practices.

DETAILED DESCRIPTION:
This study investigates the absorption efficiency of enteral nutrition in patients recovering from an intensive care unit (ICU) stay. Nutritional support is critical in the recovery of ICU patients, and enteral feeding is commonly used due to its benefits in preserving gut integrity and reducing infection risks. However, there is limited data on the actual absorption of nutrients in these patients, particularly in terms of how much of the provided energy is utilized versus excreted.

The primary focus of this study is to quantify the caloric intake and the caloric content of excreted stool to determine the efficiency of nutrient absorption in post-ICU patients. This will be done using bomb calorimetry, which measures the energy content in stool samples, and indirect calorimetry to assess the patients' resting energy expenditure (REE).

The study design is prospective, interventional, and single-center, involving 20 post-ICU patients who meet the inclusion criteria. Detailed tracking of caloric intake, including both enteral feeding and supplemental infusion calories, will be performed daily. Stool samples will be collected for three days, with the nonabsorbable blue dye marker method used to track the specific stool produced during this period. These stool samples will be freeze-dried, formed into pellets, and analyzed using the Parr 6200 Isoperibol Calorimeter to measure their energy content.

The secondary objective is to evaluate the sustainability of enteral feeding practices by assessing the amount of waste generated, such as unused nutritional formulas and tubing. This includes quantifying food waste in the hospital, focusing on nutrition that is not consumed, absorbed, or excreted.

By understanding the actual energy absorption in ICU survivors, this study aims to provide insights that will optimize nutritional strategies, improve patient recovery, and contribute to cost-effective, environmentally sustainable healthcare practices.

ELIGIBILITY:
Inclusion Criteria:

* age of 18 years or older
* minimum ICU stay of 7 days
* fully dependent on enteral feeding (nasogastric or PEG-tube)
* ability of the patient or representative to understand and sign written informed consent in Dutch, French or English

Exclusion Criteria:

* known inflammatory bowel disease
* known malabsorptive gastrointestinal disease
* history of small bowel resection
* concomitant use of serotoninergic or sympathomimetic medications (oa. setrone, tryptans, antidepressants, methylphenidate, monoamine oxidase inhibitors, tramadol)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
caloric absorption efficiency | From screening to study completion for the patient, on average 3 days
  the caloric intake from enteral feeding will be compared with the caloric content of the excreted stool. The difference between these two values will provide an estimate of how efficiently the body absorbs the administered nutrients.
Resting Energy Expenditure (REE) | From screening to study completion for the patient, on average 3 days
  The study will measure the resting energy expenditure of post-ICU patients using indirect calorimetry, which provides a real-time measure of the patients' basal metabolic rate and energy needs.

SECONDARY OUTCOMES:
Nutrient Absorption Efficiency | From screening to study completion for the patient, on average 3 days
  The proportion of the enteral nutrition that is absorbed by the patient will be compared to the total amount administered. A higher absorption efficiency would suggest less wasted nutrition and better utilization of the enteral feeding.
Waste Generation from Enteral Feeding Solutions and Tubing | From screening to study completion for the patient, on average 3 days
  The study will evaluate the quantity of waste produced from the daily replacement of enteral feeding solutions and tubing. This measure will provide insight into the sustainability impact of current practices and how much material is being discarded in hospital settings.
Overall Food Waste in Hospitals | From screening to study completion for the patient, on average 3 days
  The study will quantify the amount of enteral nutrition that is not consumed, absorbed, or excreted. This includes any nutrition that is wasted due to feeding inefficiencies or patient non-consumption.

CONTACTS AND LOCATIONS:
Locations (2):
- Belgium (2):
  - UZ Brussel, Brussels
  - UZ Brussel, Jette

IPD SHARING:
Plan to Share IPD: Undecided